CLINICAL TRIAL: NCT06129617
Title: Prospective Randomized Controlled Trial for Protein-bound Toxins Removal With Intermittent ADVOS vs. Hemodialysis Treatment in Non-intensive Care Patients With Pre-existing Liver Dysfunction and Indication for Extracorporeal Renal Support. The ADVOMITTENT Study
Brief Title: Intermittent ADVOS vs. Hemodialysis in Non-intensive Care Patients With Liver Dysfunction
Acronym: ADVOMITTENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Mainz (Other)
Collaborators: ADVITOS GmbH München (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Julia Weinmann-Menke, Head of nephrology and kidney transplantation, University Medical Center Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVOMITTENT
Record Dates: First submitted 2023-06-21; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Liver Cirrhosis; Kidney Failure, Acute; Kidney Replacement; Multi Organ Failure
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury; Multiple Organ Failure | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodialysis (Active Comparator): Patients receiving hemodialysis therapy mit Fresenius 5008
  Interventions: Device: Hemodialysis
- ADVOS (Experimental): Patients receiving ADVOS therapy with ADVOS multi
  Interventions: Device: ADVOS

INTERVENTIONS:
Device: Hemodialysis — 5 treatments with hemodialysis on day 1, 2, 3, 5 and 7
  Arms: Hemodialysis
Device: ADVOS — 5 treatments with ADVOS on day 1, 2, 3, 5 and 7
  Arms: ADVOS

SUMMARY:
In the planned randomized controlled prospective pilot study, we aim to evaluate ADVOS compared with conventional hemodialysis regarding the elimination of protein-bound toxins in patients with therapy-refractory hepatorenal syndrome.

The study will be performed in a regular non-ICU ward with a large experience in the use of the ADVOS therapy.

DETAILED DESCRIPTION:
Acute on chronic liver failure (ACLF) is a syndrome in patients with liver cirrhosis characterized by acute hepatic decompensation (i.e., jaundice, ascites, hepatic encephalopathy, bacterial infection, or gastrointestinal bleeding) and single or multi-organ failure, resulting in increased mortality. The European Association for the Study of the Liver (EASL) has established the Chronic Liver Failure (CLIF) consortium, which has developed a score for risk stratification and prognosis estimation, the CLIF-C ACLF score. Based on the CANONIC study, the CLIF consortium has developed a simplified CLIF Consortium Organ Failure Score (CLIF-C OFs), which includes liver, kidney, and lung function, hepatic encephalopathy, coagulation, and hemodynamics. Considering two other mortality factors (age and leukocyte count), the CLIF-C ACLF score was defined. The score has a higher predictive value for 28- and 90-day mortality than the Model of End Stage Liver Disease (MELD), MELD-Na, or Child-Turcotte-Pugh score.

Therapeutic options are limited and aim to address specific organ complications. In most cases, due to progressive renal insufficiency as part of hepatorenal syndrome, renal replacement therapy is if indicated. The only potential cure is liver transplantation.

There is some evidence that extracorporeal liver support can help a patient until liver transplantation or restoration of organ function. The Advanced Organ Support (ADVOS) system (ADVITOS GmbH, Munich, Germany) is an albumin-based advanced hemodialysis procedure, which can support the liver. The principles of conventional renal replacement therapy for the elimination of water-soluble substances are combined with the elimination of protein-bound substances by recirculating a dialysate containing 200 ml of human albumin. This procedure is typically used as continuous treatment in an intensive care setting. However, the investigators have already investigated the possibility of ADVOS as an intermittent procedure in patients with ACLF on a regular ward in a retrospective study.

To the best of knowledge of the investigators, there are currently no randomized studies comparing the elimination of protein-bound toxins between ADVOS and hemodialysis. Nevertheless, based on the investigators clinical experience, the investigators hypothesize that treatment with ADVOS may confer advantages over hemodialysis. Therefore, the objective of this study is to assess the effectiveness of ADVOS in comparison to hemodialysis for the treatment of patients with therapy-refractory hepatorenal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Capacity of the patient to give consent
* Pre-existing liver disease in the sense of an ACLF with HRS
* Age >18 years
* Patient of the University Medical Center Mainz
* Bilirubin level ≥ 4 mg/dl
* Indication for renal replacement procedure is based on STARRT-AKI criteria (serum potassium ≥ 6 mmol/l in two independent blood samples; serum pH of 7.2 or less or serum bicarbonate of 12 mmol/l or less; respiratory failure secondary to volume excess)

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Contraindications for ADVOS therapy
* Already started renal replacement therapy
* Contraindication for citrate anticoagulation
* Use of vasopressors and MAD ≤ 50 mmHg.
* Terminal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
course of total bilirubin in patients blood | Within 6 hours before first treatment and within 2 hours after every treatment session
  measurement of concentration of total bilirubin in serum of patients in mg/dl

SECONDARY OUTCOMES:
course of uremia toxins in patients blood | Within 6 hours before first treatment and within 2 hours after every treatment session
  measurement of blood urea nitrogen in serum of patients in mg/dl
course of bile acids | Within 6 hours before first treatment and within 2 hours after every treatment session
  measurement of bile acids in serum of patients in mg/dl
evaluation of safety of ADVOS versus hemodialysis | during the five interventions
  Rate of complications during procedure (for example hypotension, electrolyte disorders etc.)
Quality of life raised in a standardized questionnaire | baseline before intervention and on days 28, 90, 180
  We will use the WHOQOL-BREF-questionnaire with 26 questions and values from 1 to 5; 1 being the lowes value and 5 the highest value
number of days in hospital during the intervention | admission in our department till discharge from our deparment
  we will measure the number of days in the hospital during the intervention from admission to our department until discharge from our department
course of pO2 | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the pO2 (in mmHg) in a blood sample with blood gas system (ABL800 FLEX Plus)
course of pCO2 | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the pCO2 (in mmHg) in a blood sample with blood gas system (ABL800 FLEX Plus)
course of base excess | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the base excess (mmol/l) in a blood sample with blood gas system (ABL800 FLEX Plus)
course of pH | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the pH in a blood sample with blood gas system (ABL800 FLEX Plus)
course of standard bicarbonat concentration | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the standard bicarbonat concentration (mmol/l) in a blood sample with blood gas system (ABL800 FLEX Plus)
course of potassium | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the potassium (mmol/l) in a blood sample with blood gas system (ABL800 FLEX Plus)
course of sodium | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the sodium (mmol/l) in a blood sample with blood gas system (ABL800 FLEX Plus)
course of ionised calcium | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the ionised calcium (mmol/l) in a blood sample with blood gas system (ABL800 FLEX Plus)
course of bilirubin | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the bilirubin (in mg/dl) in a blood sample
course of INR | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the INR in a blood sample
course of albumin | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the albumin (in g/l) in a blood sample
course of kidney function | Within 6 hours before first treatment and within 2 hours after every treatment session
  we will measure the kreatinine (in mg/dl) in a blood sample
course of MELD | Within 6 hours before first treatment and within 2 hours after 5 treatments
  MELD = Model for End-stage Liver Disease (6-40, Higher numbers indicate increased mortality)
course of CLIF-C ACLF score | Within 6 hours before first treatment and within 2 hours after 5 treatments
  CLIF-C ACLF Score = Chronich Liver failure Consortium acute on chronic liver failure score (6-15, higher numbers indicate increased mortality)
course of hepatic encephalopathy | Within 6 hours before first treatment and within 2 hours after every treatment session
  an experienced clinician will determine the grade of the hepatic encephalopathy using the west haven criteria (grade 1 till grade 4, "grade 1" beeing the lowest value und "grade 4" beeing the highest value)
mortality | 28, 90 and 180 days.
elimination of blood urea nitrogen | Within 6 hours before first treatment and within 2 hours after every treatment session
  We will measure the Blood urea nitrogen (mg/dl) in a blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Julia Weinmann-Menke, Prof., Principal Investigator — Principal Investigator
Locations (1):
- UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz I. Medizinische Klinik und Poliklinik, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Undecided